CLINICAL TRIAL: NCT03220997
Title: Do Preoperative Carbohydrate Drinks Prevent Preoperative Catabolism in Mothers Undergoing Elective Caesarean Section? A Randomised Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Obstetric Anaesthetists' Association United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GN16OG711
Record Dates: First submitted 2017-06-06; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Starvation; Caesarean Section
Keywords: Sequela; Ketosis
MeSH Terms: conditions — Starvation; Ketosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Research midwives will attend consent, randomise, collect baseline data and provide the accompanying information and carbohydrate sachets to subjects. The research fellows will be blinded but will collect the data for participants. The research midwives will complete study compliance. To achieve this, participants will bring to ward a completed compliance form ( given at randomisation) in a sealed envelope this will ensure the research investigators remain blinded during their pre op assessments and data collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Mothers will be given six sachets of carbohydrate powder to be mixed in water . Instructions will be given to have two sachets in 800ml water at 10pm the night before and one sachet in 400ml water at 6 am on the morning of surgery. The order of the list will be decided at 8.45am on the morning of surgery by the surgical team. Mothers scheduled to have surgery later than 11am will be given a further sachet at 9.30am. Mothers scheduled for surgery after 1pm will be given a sachet at 9am and 11am.
  Interventions: Dietary Supplement: Vitaflow Preload
- Standard Care (No Intervention): Standard fasting instructions will given to mother:
  Food until midnight before surgery 800ml water at 10pm night before surgery 400ml water at 6 am morning of surgery The order of the list will be decided at 8.45am on the morning of surgery by the surgical team.
  Mothers scheduled to have surgery later than 11am will be given a further 400ml water at 9.30am. Mothers scheduled for surgery after 1pm will be given 400ml water at 9am and 11am.

INTERVENTIONS:
Dietary Supplement: Vitaflow Preload — Carbohydrate loading drink
  Arms: Interventional

SUMMARY:
The primary aim of this randomised control trial is to assess the impact of pre-operative carbohydrate loading on the incidence of urinary ketone bodies when compared to standard care in elective caesarean section. Half of the participants will receive pre-operative carbohydrates and the other half will receive standard care.

DETAILED DESCRIPTION:
Patients requiring general anaesthetic for surgical procedures are asked to stop eating and drinking for several hours before the procedure. This is due to concerns that such patients are at risk of lung damage caused by stomach contents entering their lungs while they are asleep (aspiration of gastric contents).

However, fasting patients for long periods of time can lower their ability to heal well and slow their recovery from surgery. Fasting increases anxiety levels and leads to poor patient satisfaction with the care received.

Recent studies have showed that allowing patients to drink clear, easily absorbed sugar rich liquids (carbohydrate drinks) until two hours prior to their anaesthetic does not expose them to extra risks while preventing the deleterious effects of starvation.

Carbohydrate drinks with a few other measures aimed at facilitating early recovery after surgeries are collectively termed Enhanced recovery after surgery (ERAS). The benefits and safety of enhanced recovery have been demonstrated in patients undergoing major bowel surgery and have been widely adopted. However, so far, no studies have been conducted to determine if these results apply to mothers undergoing planned caesarean sections. We hope to address this gap in the knowledge with our proposed study.

All mothers undergoing a planned caesarean section in the Princess Royal Maternity (PRM) will be invited to participate. Mothers will be divided into two groups. One group will receive standard care and the other group will receive a carbohydrate drink in addition to standard care. Information collected from the groups will be compared to evaluate the expected benefits and risks. The study will continue until the target sample size of 100 mothers in each of the two study groups is reached.

ELIGIBILITY:
Inclusion Criteria:

* Mother scheduled for elective caesarean delivery at the Princess Royal Maternity Unit, Glasgow.

Exclusion Criteria:

* Patient refusal
* Severe oesophageal reflux disease (persistent daytime and night-time reflux in association with documented structural damage i.e. Barrett's Oesophagus.)
* Diabetes mellitus requiring treatment beyond dietary modulation
* Unable to consent
* Patients undergoing general anaesthetic should be excluded from the study.
* Anticipated complex caesarean section patients.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of urine ketone body levels at catheterisation prior to elective caesarean delivery. | From insertion of urinary catheter until 5 minutes post urinary catherisation
  After bladder catheterisation, urine will be tested for ketone bodies (Ketostix, Bayer)

SECONDARY OUTCOMES:
Preoperative thirst | On arrival to theatre - 5 minutes duration for questioning
  Assessed via visual analogue scale
Preoperative hand grip strength | On arrival to theatre and immediately prior to discharge from recovery room - 4 hour duration
  Dominant hand grip strength measures with dynamometer
Length of hospital stay | From admission to hospital until the date of discharge or date of death from any cause, whichever came first, assessed up to two weeks duration
  Measured length of stay between hospital admission and discharge home

OTHER OUTCOMES:
Incidence of aspiration of gastric contents under general anaesthesia | From date of randomization until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to two weeks duration
  Inhalation of gastric contents

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Obstetric Anaesthetists' Association (2012). GENERAL ANAESTHETIC FOR UNPLANNED CAESAREAN SECTION (CS) INFORMATON CARD. http://www.labourpains.com/assets/_managed/editor/File/Info%20for%20Mothers/GA%20for%20unplanned%20CS/GA_Unplanned_CS.pdf.pdf accessed 23/04/15.
- [Background] Clark, A & Agaram, R. (2014) Too fast? Ketonuria as a marker of prolonged fasting in elective caesarean section. International Journal of Obstetric Anaesthesia 23, Supplement 1, S1-S62.
- [Background] Metzger BE, Ravnikar V, Vileisis RA, Freinkel N. "Accelerated starvation" and the skipped breakfast in late normal pregnancy. Lancet. 1982 Mar 13;1(8272):588-92. doi: 10.1016/s0140-6736(82)91750-0. PMID 6121184
- [Background] Agarwal A, Chari P, Singh H. Fluid deprivation before operation. The effect of a small drink. Anaesthesia. 1989 Aug;44(8):632-4. doi: 10.1111/j.1365-2044.1989.tb13581.x. PMID 2782569
- [Background] Lucas DN, Gough KL. Enhanced recovery in obstetrics--a new frontier? Int J Obstet Anesth. 2013 Apr;22(2):92-5. doi: 10.1016/j.ijoa.2013.02.001. Epub 2013 Mar 9. No abstract available. PMID 23477889
- [Background] Wong CA, Loffredi M, Ganchiff JN, Zhao J, Wang Z, Avram MJ. Gastric emptying of water in term pregnancy. Anesthesiology. 2002 Jun;96(6):1395-400. doi: 10.1097/00000542-200206000-00019. PMID 12170052
- [Background] Wong CA, McCarthy RJ, Fitzgerald PC, Raikoff K, Avram MJ. Gastric emptying of water in obese pregnant women at term. Anesth Analg. 2007 Sep;105(3):751-5. doi: 10.1213/01.ane.0000278136.98611.d6. PMID 17717235
- [Background] Smith I, Kranke P, Murat I, Smith A, O'Sullivan G, Soreide E, Spies C, in't Veld B; European Society of Anaesthesiology. Perioperative fasting in adults and children: guidelines from the European Society of Anaesthesiology. Eur J Anaesthesiol. 2011 Aug;28(8):556-69. doi: 10.1097/EJA.0b013e3283495ba1. PMID 21712716
- [Background] Gustafsson UO, Scott MJ, Schwenk W, Demartines N, Roulin D, Francis N, McNaught CE, Macfie J, Liberman AS, Soop M, Hill A, Kennedy RH, Lobo DN, Fearon K, Ljungqvist O; Enhanced Recovery After Surgery (ERAS) Society, for Perioperative Care; European Society for Clinical Nutrition and Metabolism (ESPEN); International Association for Surgical Metabolism and Nutrition (IASMEN). Guidelines for perioperative care in elective colonic surgery: Enhanced Recovery After Surgery (ERAS((R))) Society recommendations. World J Surg. 2013 Feb;37(2):259-84. doi: 10.1007/s00268-012-1772-0. No abstract available. PMID 23052794
- [Background] Nygren J, Thorell A, Jacobsson H, Larsson S, Schnell PO, Hylen L, Ljungqvist O. Preoperative gastric emptying. Effects of anxiety and oral carbohydrate administration. Ann Surg. 1995 Dec;222(6):728-34. doi: 10.1097/00000658-199512000-00006. PMID 8526579
- [Background] Gustafsson UO, Hausel J, Thorell A, Ljungqvist O, Soop M, Nygren J; Enhanced Recovery After Surgery Study Group. Adherence to the enhanced recovery after surgery protocol and outcomes after colorectal cancer surgery. Arch Surg. 2011 May;146(5):571-7. doi: 10.1001/archsurg.2010.309. Epub 2011 Jan 17. PMID 21242424
- [Background] Clark A, Litchfield K, Hannah S, Love C, Slade K, Lake K, Agaram R. Pre-operative carbohydrate loading prior to elective caesarean delivery: a randomised controlled trial. Int J Obstet Anesth. 2021 Feb;45:21-27. doi: 10.1016/j.ijoa.2020.10.008. Epub 2020 Oct 18. PMID 33277162
- [Background] Neufer PD, Costill DL, Flynn MG, Kirwan JP, Mitchell JB, Houmard J. Improvements in exercise performance: effects of carbohydrate feedings and diet. J Appl Physiol (1985). 1987 Mar;62(3):983-8. doi: 10.1152/jappl.1987.62.3.983. PMID 3571097
- [Background] Gustafsson UO, Nygren J, Thorell A, Soop M, Hellstrom PM, Ljungqvist O, Hagstrom-Toft E. Pre-operative carbohydrate loading may be used in type 2 diabetes patients. Acta Anaesthesiol Scand. 2008 Aug;52(7):946-51. doi: 10.1111/j.1399-6576.2008.01599.x. Epub 2008 Mar 7. PMID 18331374
- [Result] Scott MJ, Fawcett WJ. Oral carbohydrate preload drink for major surgery - the first steps from famine to feast. Anaesthesia. 2014 Dec;69(12):1308-13. doi: 10.1111/anae.12921. Epub 2014 Oct 23. No abstract available. PMID 25346490